CLINICAL TRIAL: NCT01680822
Title: Treatment Outcomes in Patient With Nontuberculous Mycobacterial Disease in the University of Illinois Hospital & Health Sciences System
Brief Title: Treatment Outcomes in Patient With Nontuberculous Mycobacterial Disease
Status: Terminated | Type: Observational
Why Stopped: PI left institution, not able to contact; data destroyed
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Erin Vidra, Fellow, Pulmonary and Critical Care, University of Illinois at Chicago
Other Study IDs: 2012-0662; UIC (Other: University of Illinois at Chicago)
Record Dates: First submitted 2012-08-31; First posted 2012-09-07 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Nontuberculous Mycobacterial Disease; Atypical Mycobacterium Infections
Keywords: Nontuberculous, Atypical, Mycobacterial
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NTM patient: confirmed NTM patient

SUMMARY:
Little is known about the disease caused by the nontuberculous or environmental mycobacteria (NTM) and only limited data are available showing treatment outcome. This project will study the patients with nontuberculous mycobacterial (NTM) diseases in the University of Illinois Hospital & Health Sciences System (UIMC). The aim of study is finding treatment outcome and risk factors that are associated with treatment failure in NTM patients. This is a retrospective, observational study for collecting data on patients with NTM in UIMC. The study initially involves populating the study of NTM patients seen at UIMC during the study period. This will add our knowledge about current treatment outcome of patients with NTM diseases and will be of interest to physicians, and public health authorities.

DETAILED DESCRIPTION:
The study focuses on collecting all mycobacterial data, clinical assessment and clinical outcomes of patients. Data collection includes demographic characteristics, medical history, clinical procedures relative to the treatment of NTM, respiratory symptoms and signs, pulmonary function tests if applicable, imaging parameters, diagnostic tests, mycobacterial smear, culture, or possible susceptibility, therapies and outcome. The study will be updated with clinical outcomes (e.g., hospitalization, surgery relative NTM, and death) during study period. The data will be collected from 1/1/2001 to 12/30/ 2011.

The confirmed NTM patient will be defined with ATS guideline for NTM as:

Clinical: Pulmonary symptoms, nodular or cavitary opacities on chest radiograph, or an HRCT scan that shows multifocal bronchiectasis with multiple small nodules and 2. appropriate exclusion of other diagnoses.

Microbiologic: Positive culture results from at least two separate expectorated sputum samples. (If the results from the initial sputum samples are nondiagnostic, we will consider repeat sputum AFB smears and cultures.) Or positive culture results from at least one bronchial wash or lavage. Or transbronchial or other lung biopsy with mycobacterial histopathologic features (granulomatous inflammation or AFB) and positive culture for NTM or biopsy showing mycobacterial histopathologic features (granulomatous inflammation or AFB) and one or more sputum or bronchial washings that are culture positive for NTM.

OBJECTIVES

1. To determine prevalence of culture-confirmed NTM infection in the UIMC in a ten- year period
2. To determine the prevalence of NTM disease based on ATS case definition the UIMC in a ten- year period
3. To determine treatment outcome of NTM disease in the UIMC in a ten- year period
4. To find the risk factors associated with treatment failure of patients with NTM diseases

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 year or older with at least one culture-confirmed NTM.

Exclusion Criteria:

* All patients aged younger than 18 years old.
* No individuals are excluded from study based on, race, ethnicity, gender, or HIV status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were seeking or receiving medical care for NTM disease at UIC Medical Center that satisfy the inclusion and exclusion criteria of study are eligible to participation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Mirsaeidi, MD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Tabarsi P, Baghaei P, Farnia P, Mansouri N, Chitsaz E, Sheikholeslam F, Marjani M, Rouhani N, Mirsaeidi M, Alipanah N, Amiri M, Masjedi MR, Mansouri D. Nontuberculous mycobacteria among patients who are suspected for multidrug-resistant tuberculosis-need for earlier identification of nontuberculosis mycobacteria. Am J Med Sci. 2009 Mar;337(3):182-4. doi: 10.1097/maj.0b013e318185d32f. PMID 19301453
- [Background] Mirsaeidi M, Hadid W, Ericsoussi B, Rodgers D, Sadikot RT. Non-tuberculous mycobacterial disease is common in patients with non-cystic fibrosis bronchiectasis. Int J Infect Dis. 2013 Nov;17(11):e1000-4. doi: 10.1016/j.ijid.2013.03.018. Epub 2013 May 16. PMID 23683809
- [Background] Mirsaeidi M, Farshidpour M, Ebrahimi G, Aliberti S, Falkinham JO 3rd. Management of nontuberculous mycobacterial infection in the elderly. Eur J Intern Med. 2014 Apr;25(4):356-63. doi: 10.1016/j.ejim.2014.03.008. Epub 2014 Mar 29. PMID 24685313
- [Background] Mirsaeidi M, Machado RF, Garcia JG, Schraufnagel DE. Nontuberculous mycobacterial disease mortality in the United States, 1999-2010: a population-based comparative study. PLoS One. 2014 Mar 14;9(3):e91879. doi: 10.1371/journal.pone.0091879. eCollection 2014. PMID 24632814